## **ICF**

## **MOSART-study**

Neurotoxic adverse effects of morphine and oxycodone in continuous subcutaneous infusion for treatment of pain in terminal patients with diminished renal function: a Randomized Controlled Trial.

Version number: 2, date 2017.08.18

# Proefpersoneninformatie voor deelname aan medisch-wetenschappelijk onderzoek

#### **MOSART-studie**

Een onderzoek naar verschillen in bijwerkingen tussen morfine en oxycodon bij continue toediening voor behandeling van pijn bij personen in de stervensfase.

Officiële titel: Neurotoxische bijwerkingen van morfine en oxycodon voor continue subcutane infusie ter behandeling van pijn bij terminale patiënten met een verminderde nierfunctie: een Randomized Controlled Trial.

## Inleiding

Geachte heer/mevrouw,

Wij vragen u om mee te doen aan een medisch-wetenschappelijk onderzoek. Meedoen is vrijwillig. Om mee te doen is wel uw schriftelijke toestemming nodig.

U ontvangt deze brief omdat uw behandelend arts heeft vastgesteld dat continue toediening van een opioïd (een sterke pijnstiller) nodig is om pijn in uw laatste levensfase te behandelen.

Voordat u beslist of u wilt meedoen aan dit onderzoek, krijgt u uitleg over wat het onderzoek inhoudt. Lees deze informatie rustig door en vraag de onderzoeker om uitleg als u vragen heeft. U kunt ook de onafhankelijke deskundige, die aan het eind van deze brief genoemd wordt, om aanvullende informatie vragen. En u kunt er ook over praten met uw partner, vrienden of familie.

Verdere informatie over meedoen aan zo'n onderzoek staat in de bijgevoegde brochure 'Medisch-wetenschappelijk onderzoek'.

## 1. Algemene informatie

Dit onderzoek is opgezet door het Expertisecentrum Palliatieve Zorg van het Maastricht Universitair Medisch Centrum en wordt gedaan door artsen en onderzoekers in verschillende verpleeghuizen en hospices. Voor dit onderzoek zijn in totaal 234 proefpersonen nodig.

Dit onderzoek wordt mede mogelijk gemaakt door een subsidie van ZonMw en cofinanciering door Envida en het Maastricht Universitair Medisch Centrum.

De medisch ethische toetsingscommissie van het azM/UM (METC azM/UM) heeft dit onderzoek goedgekeurd. Algemene informatie over de toetsing van onderzoek vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

#### 2. Doel van het onderzoek

Het doel van dit onderzoek is het vergelijken van bepaalde bijwerkingen bij het continu toedienen van morfine of oxycodon voor pijnbestrijding bij patiënten in de laatste levensfase met een verminderde nierfunctie.

## 3. Achtergrond van het onderzoek

In de laatste levensfase komt pijn vaak voor. De 'morfine-pomp' is een veel gebruikte behandeling voor deze pijn. Hierbij wordt continu een hoeveelheid morfine toegediend via een klein onderhuids naaldje (dit noemen we subcutane infusie). Een andere mogelijkheid is dat om de vier uur een vergelijkbare hoeveelheid morfine via dit onderhuidse naaldje wordt toegediend. Beide methodes werken even goed.

Het is echter de vraag of morfine wel het meest geschikte middel is in deze situatie. Door achteruitgang van lichaamsfuncties in deze laatste levensfase, waaronder vermindering van de nierfunctie, kunnen afbraakproducten van morfine zich namelijk gaan opstapelen in het lichaam. We vermoeden dat door deze opstapeling van afbraakproducten mogelijk bijwerkingen zouden kunnen ontstaan, zoals onrust en/of verwardheid (in medische termen wordt dit een delier genoemd) of zelfs toegenomen pijnbeleving. Dit zou dan kunnen leiden tot een sterfbed met toenemende onrust en/of pijn, terwijl we juist het tegenovergestelde proberen te bereiken.

Oxycodon is een middel dat vergelijkbaar is met morfine. Het zijn beide sterke pijnstillers, die we opioïden noemen. Oxycodon wordt net als morfine al langdurig in de praktijk toegepast en heeft geen nadelen ten opzichte van morfine. De keuze voor één van beide middelen berust in de praktijk vaak op de persoonlijke voorkeur van de arts. Oxycodon heeft echter minder opstapelende afbraakproducten dan morfine. We denken dat hierdoor in theorie bij oxycodon minder van de genoemde vervelende bijwerkingen zouden kunnen optreden.

Dat is echter op dit moment alleen nog maar een theorie, die nog nooit eerder goed is onderzocht. Het is hierdoor nog onbekend of oxycodon in de praktijk ook echt minder van de genoemde bijwerkingen geeft dan morfine. Dat willen we met dit onderzoek gaan vergelijken. Met de uitkomsten van dit onderzoek zouden we een belangrijke bijdrage kunnen leveren aan het verbeteren van de kwaliteit van zorg voor mensen in de laatste levensfase.

#### 4. Wat meedoen inhoudt

Deelname aan het onderzoek duurt net zo lang als uw behandeld arts nodig vindt dat u de pijnstiller toegediend krijgt. In de praktijk is dit vrijwel altijd tot aan uw overlijden.

#### Geschiktheidsonderzoek

Om deel te kunnen nemen aan dit onderzoek hebben wij uiteraard uw toestemming nodig. Hiervoor dient het toestemmingsformulier door u ondertekent te worden. Als u uw toestemming heeft gegeven, zullen we vervolgens eerst bepalen of u ook daadwerkelijk geschikt bent om mee te doen. Hiervoor hebben we uw medische gegevens nodig van uw behandelend arts. Daarnaast zullen we bij het eerste bezoek eenmalig bloed bij u moeten prikken. Dat is nodig om uw nierfunctie te bepalen. Als uit het bloedonderzoek blijkt dat uw nierfunctie niet verminderd is, stopt op dat moment voor u de verdere deelname aan het onderzoek.

Als u dit niet wilt, kunt u niet meedoen aan dit onderzoek.

#### Behandeling

De ene helft van de studiedeelnemers krijgt morfine, de andere helft oxycodon. Loting bepaalt welke van deze twee pijnstillers u krijgt. Dit middel zal na de loting gewoon door uw eigen arts worden voorgeschreven. U blijft verder ook volledig de normale zorg van uw eigen arts ontvangen, zoals u dat anders ook zou krijgen.

De onderzoeksverpleegkundige die gedurende het onderzoek steeds bij u langs komt, weet niet in welke groep u zit. Zo wordt hij/zij niet beïnvloed bij het uitvoeren van de metingen. Het is dan ook belangrijk dat u hem/haar niet vertelt welke van de twee pijnstillers u krijgt.

Algemene informatie hierover vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

#### Bezoeken en metingen

Wij komen u bezoeken in uw eigen kamer in het verpleeghuis of hospice waar u verblijft. U hoeft dus zelf niet te reizen. Deze bezoeken worden uitgevoerd door (één van) onze onderzoeksverpleegkundigen.

Bij het eerste bezoek zal de onderzoeksverpleegkundige eenmalig één buisjes bloed bij u afnemen. Dit is om uw nierfunctie te bepalen.

Vervolgens zal de onderzoeksverpleegkundige u drie keer per week bezoeken. Een bezoek duurt ongeveer tien minuten. Er zal dan het volgende gebeuren:

- Wij vragen u om aan te geven hoeveel pijn u heeft. Als u niet (meer) in staat bent om dit aan te geven, kijken wij of we kenmerken van pijn bij u kunnen zien.
- Wij strijken kort met een watje over uw onderarmen en vragen u of dit pijnlijk aanvoelt. Als u niet (meer) in staat bent om dit aan te geven, kijken wij of we bij u kenmerken van een pijnlijke reactie kunnen zien.
- Wij laten kort een scherpe naald op uw onderarmen rusten (zonder u te prikken uiteraard) en vragen u of dit pijnlijk aanvoelde. Als u niet (meer) in staat bent om dit aan te geven, kijken wij of we bij u kenmerken van een pijnlijke reactie kunnen zien.

Daarnaast zal de onderzoeksverpleegkundige bij elk bezoek de volgende informatie verzamelen bij het verzorgend personeel van uw afdeling:

- De medicatie die u op dat moment gebruikt.
- Of zij tekenen van een delier (onrust/verwardheid) bij u hebben waargenomen.
- Of zij nog andere bijwerkingen bij u hebben waargenomen.

Na uw overlijden zouden wij graag een naaste van u, die veel bij u aanwezig was in de periode rond uw overlijden, telefonisch willen benaderen voor een interview door de onderzoeker over hoe deze persoon deze periode heeft ervaren. Dit telefonisch interview mag alleen plaatsvinden als zowel u, als uw naaste hier toestemming voor geven.

#### 5. Wat wordt er van u verwacht

Om het onderzoek goed te doen verlopen, is het belangrijk dat u zich aan de volgende afspraken houdt.

De afspraken zijn dat u:

- het onderzoeksmiddel toe laat dienen volgens het voorschrift van uw arts.
- niet ook nog aan een ander medisch-wetenschappelijk onderzoek meedoet.
- afspraken voor bezoeken aan u respecteert.
- de onderzoeksverpleegkundige(n) niet vertelt welke van de twee pijnstillers u krijgt.

#### 6. Mogelijke bijwerkingen

De onderzoeksmiddelen morfine en oxycodon kunnen bijwerkingen geven.

Deze bijwerkingen komen vaak voor (bij 1 op de 10 mensen of meer):

- Obstipatie. Uw arts kan u hiervoor een laxeermiddel voorschrijven.
- Misselijkheid en braken. Dit verdwijnt meestal na een paar dagen. Uw arts kan u tijdelijk een middel tegen de misselijkheid voorschrijven.
- Slaperigheid of sufheid. Dit verdwijnt meestal na een paar dagen.

- Droge mond. Uw arts kan u middelen voorschrijven die deze klachten kunnen verminderen.

Deze bijwerkingen komen voor, maar niet zo vaak:

- Jeuk. Uw arts kan u een middel voorschrijven dat deze klachten kan verminderen.
- Onvolledige blaaslediging (blaasretentie). Een blaaskatheter kan de klachten hiervan wegnemen.

De onderzoeksmiddelen kunnen ook bijwerkingen hebben die nog onbekend zijn.

Meer informatie over oxycodon en morfine staat in de bijsluiters. Doet u mee aan het onderzoek? Dan kunt u uw behandelend arts hierom vragen.

#### Metingen

Een bloedafname kan pijn doen of een bloeduitstorting geven.

Het strijken met een watje over de huid of het plaatsen van een scherpe naald op de huid kan mogelijk kortdurend een pijnlijke reactie oproepen bij het uitvoeren hiervan.

## 7. Mogelijke voor- en nadelen

Het is belangrijk dat u de mogelijke voor- en nadelen goed afweegt voordat u besluit mee te doen.

## Voordelen

Wanneer u door loting in de morfine-groep wordt ingedeeld, heeft u zelf geen voordeel van meedoen aan dit onderzoek. Uw deelname kan wel bijdragen aan meer kennis over de behandeling van pijn in de terminale fase.

Wanneer u door loting in de oxycodon-groep wordt ingedeeld, kan de kans kleiner worden dat bij u onrust/verwardheid (een delier) of een toegenomen pijnbeleving optreedt, maar zeker is dat niet.

## Nadelen

Een nadeel van meedoen aan het onderzoek kan zijn dat u mogelijk ongemakken ondervindt van de metingen in het onderzoek.

Deelname aan het onderzoek betekent ook:

- dat u in uw laatste levensperiode drie maal per week bezoek krijgt van een 'vreemde' onderzoeksverpleegkundige;
- dat u tijdens dit bezoek 5 tot 10 minuten tijd kwijt bent;
- dat u afspraken heeft waaraan u zich moet houden.

Al deze zaken zijn hiervoor onder punt 4, 5 en 6 beschreven. Uiteraard zullen wij ons maximaal inspannen om de overlast voor u tot een minimum te beperken.

## 8. Als u niet wilt meedoen of wilt stoppen met het onderzoek

U beslist zelf of u meedoet aan het onderzoek. Deelname is vrijwillig.

Als u niet wilt meedoen, wordt u op de gebruikelijke manier behandeld voor uw pijn. Het feit dat u voor deelname aan dit onderzoek in aanmerking komt, betekent dat uw behandelend arts al heeft vastgesteld dat deze behandeling het beste kan plaatsvinden met continue toediening van een opioïd. Uw behandelend arts bepaalt dan zelf welk opioïd u toegediend krijgt.

Als u wel meedoet, kunt u zich altijd bedenken en toch stoppen, ook tijdens het onderzoek. U wordt dan weer op de gebruikelijke manier behandeld voor uw pijn. U hoeft niet te zeggen waarom u stopt. Wel moet u dit direct melden aan de onderzoeker.

De gegevens die tot dat moment zijn verzameld, worden gebruikt voor het onderzoek.

Als er nieuwe informatie over het onderzoek is die belangrijk voor u is, laat de onderzoeker dit aan u weten. U wordt dan gevraagd of u blijft meedoen.

#### 9. Einde van het onderzoek

Uw deelname aan het onderzoek stopt als

- uit het bloedonderzoek blijkt dat u geen verminderde nierfunctie heeft;
- alle bezoeken zoals beschreven onder punt 4 voorbij zijn;
- u zelf kiest om te stoppen;
- uw behandelend arts het niet langer nodig vindt dat u met een opioïd behandeld wordt;
- de onderzoeker het beter voor u vindt om te stoppen;
- uw behandelend arts het beter voor u vindt om te stoppen;
- u verhuist buiten de deelnemende instellingen;
- het Expertisecentrum Palliatieve Zorg MUMC+, ZonMw, Envida, de overheid of de beoordelende medisch ethische toetsingscommissie besluiten om het onderzoek te stoppen.

Het hele onderzoek is afgelopen als alle deelnemers zijn overleden of om de overige genoemde redenen met deelname aan het onderzoek zijn gestopt.

Morfine en oxycodon zijn gangbare middelen, die door uw eigen behandelend arts worden voorgeschreven. Wanneer u besluit dat u wilt stoppen met uw deelname aan het onderzoek blijft hierdoor de medicatie die u gebruikt heeft tijdens het onderzoek naderhand beschikbaar via uw behandelend arts. Uiteraard alleen wanneer uw behandelend arts het gebruik van

deze middelen voor u nodig acht. De onderzoeker zal met u praten over de mogelijkheden voor verdere medische zorg.

#### 10. Gebruik en bewaren van uw gegevens en lichaamsmateriaal

Voor dit onderzoek is het nodig dat uw bloed en uw medische en persoonsgegevens worden verzameld en gebruikt. Elke proefpersoon krijgt een code die op het bloedbuisje en de gegevens komt te staan. Uw naam en andere persoonsgegevens worden weggelaten.

#### Uw gegevens

Al uw gegevens blijven vertrouwelijk. Alleen de onderzoekers en de onderzoeksverpleegkundigen weten welke code u heeft. De sleutel voor de code blijft bij de onderzoeker. Ook in rapporten over het onderzoek wordt alleen die code gebruikt.

Sommige mensen mogen uw medische en persoonsgegevens inzien. Dit is om te controleren of het onderzoek goed en betrouwbaar uitgevoerd is. Algemene informatie hierover vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

Mensen die uw gegevens kunnen inzien zijn: het onderzoeksteam, een controleur die door de uitvoerder van het onderzoek is ingehuurd en de Inspectie voor de Gezondheidszorg. Zij houden uw gegevens geheim. Als u de toestemmingsverklaring ondertekent, geeft u toestemming voor het verzamelen, bewaren en inzien van uw medische en persoonsgegevens.

De onderzoeker bewaart uw gegevens 15 jaar.

#### Uw lichaamsmateriaal

Het bloed dat bij u afgenomen is, wordt door de onderzoeksverpleegkundige naar het Centraal Diagnostisch Laboratorium van het MUMC+ gebracht. Daar wordt het enkel gebruikt voor het bepalen van uw nierfunctie. Na deze bepaling wordt het bloed niet bewaard of voor andere doeleinden gebruikt.

Algemene informatie over de registratie van onderzoeken vindt u in de brochure 'Medischwetenschappelijk onderzoek'.

## 11. Verzekering voor proefpersonen

Voor iedereen die meedoet aan dit onderzoek is een verzekering afgesloten. De verzekering dekt schade door het onderzoek. Niet alle schade is gedekt. In bijlage B vindt u meer informatie over de verzekering. Daar staat ook aan wie u schade kunt melden.

#### 12. Informeren behandelend arts en apotheker

Wij sturen uw behandelend arts en apotheker van het verpleeghuis of hospice waar u verblijft altijd een brief om te laten weten dat u meedoet aan het onderzoek. Dit is voor uw eigen veiligheid. Als u dit niet goed vindt, kunt u niet meedoen aan dit onderzoek.

## 13. Geen vergoeding voor meedoen

Deelname aan dit onderzoek kost u niets. U wordt niet betaald voor het meedoen aan dit onderzoek.

## 14. Heeft u vragen?

Bij vragen kunt u contact opnemen met de onderzoeker. Voor onafhankelijk advies over meedoen aan dit onderzoek kunt u terecht bij de onafhankelijke arts. Hij weet veel over het onderzoek, maar heeft niets te maken met dit onderzoek.

Bij klachten kunt u het beste terecht bij de klachtencommissie van uw instelling. Alle gegevens vindt u in **bijlage A**: Contactgegevens.

## 15. Ondertekening toestemmingsformulier

Wanneer u voldoende bedenktijd heeft gehad, wordt u gevraagd te beslissen over deelname aan dit onderzoek. Indien u toestemming geeft, zullen wij u vragen deze op de bijbehorende toestemmingsverklaring schriftelijk te bevestigen. Door uw schriftelijke toestemming geeft u aan dat u de informatie heeft begrepen en instemt met deelname aan het onderzoek. Het handtekeningenblad overhandigt u aan uw behandelend arts. Dit zal vervolgens door de onderzoeker opgehaald en bewaard worden. U krijgt een kopie of een tweede exemplaar van deze toestemmingsverklaring.

Indien u toestemming heeft gegeven dat een naaste na uw overlijden benaderd mag worden voor een telefonisch interview, zal ook aan deze persoon gevraagd worden om een toestemmingsverklaring hiervoor te ondertekenen. Ook deze toestemmingsverklaring kan overhandigd worden aan uw behandelend arts en zal vervolgens door de onderzoeker opgehaald en bewaard worden.

Dank voor uw aandacht.

## 16. Bijlagen bij deze informatie

- A. Contactgegevens voor Envida
- B. Informatie proefpersonenverzekering
- C. Toestemmingsformulier proefpersoon
- D. Toestemmingsformulier nabestaande
- E. Brochure 'Medisch-wetenschappelijk onderzoek. Algemene informatie voor de proefpersoon' (versie mrt 2017)

## Bijlage A: contactgegevens voor Envida

Onderzoeker: Drs. M.J.M. (Mark) Martens

specialist ouderengeneeskunde, Envida

consulent palliatieve zorg, Expertisecentrum Palliatieve Zorg MUMC+

Tel.: 043 - 85093084

Onafhankelijk arts: Dr. med. M.N. (Markus) Janssen, FIPP

anesthesioloog/pijngeneeskundige MUMC+

Tel.: 043 - 3875606

Klachten: Elly Wijnen

klachtenfunctionaris Stichting Envida Tel.: 0900 - 2233440 / 06 - 23863129

E-mail: klachten@envida.nl

## Bijlage B: INFORMATIE PROEFPERSONENVERZEKERING

#### **VERZEKERINGSVERKLARING**

voor het hierna te noemen wetenschappelijk onderzoek

Titel: Neurotoxic adverse effects of morphine and oxycodone in continuous subcutaneous infusion for treatment of pain in terminal patients with diminished renal function: a Randomized Controlled Trial.

Voor iedereen die meedoet aan dit onderzoek, heeft het academisch ziekenhuis Maastricht, hierna te noemen azM, een verzekering afgesloten. De verzekering dekt schade door deelname aan het onderzoek. Dit geldt voor schade tijdens het onderzoek of binnen vier jaar na het einde ervan. Schade moet u binnen die vier jaar aan de verzekeraar hebben gemeld.

De verzekering dekt niet alle schade. Onderaan deze tekst staat in het kort welke schade niet wordt gedekt. Deze bepalingen staan in het Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen. Dit besluit staat op www.ccmo.nl, de website van de Centrale Commissie Mensgebonden Onderzoek (zie 'Bibliotheek' en dan 'Weten regelgeving').

Bij schade kunt u direct contact leggen met de verzekeraar:

De verzekeraar van het onderzoek is:

Naam: CNA Insurance Company Ltd.

Adres: World Trade Centre, Strawinskylaan 703, 1077 XX Amsterdam

Telefoonnummer: 020-5737272

Polisnummer: 10174880

Contactpersoon: Esther van Herk, Snr Claims Examiner

E-mail: Esther.VanHerk@cnaeurope.com

Telefoonnummer: 020-5737274

De verzekering biedt een dekking van ten minste € 650.000 per proefpersoon en ten minste € 5.000.000 voor het hele onderzoek (en ten minste € 7.500.000 per jaar voor alle onderzoeken van het azM).

De verzekering dekt de volgende schade niet:

- schade door een risico waarover u in de schriftelijke informatie bent ingelicht. Dit geldt niet als het risico zich ernstiger voordoet dan was voorzien of als het risico heel onwaarschijnlijk was;
- schade aan uw gezondheid die ook zou zijn ontstaan als u niet aan het onderzoek had meegedaan;
- schade door het niet (volledig) opvolgen van aanwijzingen of instructies;
- schade aan uw nakomelingen, als gevolg van een negatief effect van het onderzoek op u of uw nakomelingen;
- schade door een bestaande behandelmethode bij onderzoek naar bestaande behandelmethoden.

## Bijlage C: toestemmingsformulier proefpersoon

#### **MOSART-studie**

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn voldoende beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen of te stoppen met het onderzoek. Daarvoor hoef ik geen reden te geven.
- Ik geef toestemming voor het informeren van mijn behandelend arts en de apotheker van het verpleeghuis of hospice waar ik verblijf, dat ik meedoe aan dit onderzoek.
- Ik geef toestemming voor het opvragen van informatie bij mijn behandelend arts in het verpleeghuis of hospice waar ik verblijf over mijn medische voorgeschiedenis, huidige medische toestand en medicatiegebruik.
- Ik weet dat sommige mensen mijn gegevens kunnen inzien. Die mensen staan vermeld in deze informatiebrief.
- Ik geef toestemming voor het verzamelen en gebruiken van mijn gegevens en bloedmonster op de manier en voor de doelen die in de informatiebrief staan (zie ook sectie 4 onder geschiktheidsonderzoek).
- Ik geef toestemming om mijn gegevens op de onderzoek-locatie nog 15 jaar na dit onderzoek te bewaren.
- Ik geef toestemming om de data die dit onderzoek oplevert eventueel in de toekomst te hergebruiken voor controle of verdere analyse in het kader van wetenschappelijk onderzoek.

| - | lk geef | □ wel | |
|---|---|---|---|
| | | □ niet | |
| toestemming om na mijn overlijden de ondergenoemde persoon tele | | | noemde persoon telefonisch |
| | | te benaderen voor een interview door de onderzoeker over hoe deze | |
| | | persoon de periode rond uw overlijden heeft ervaren. Hij/zij behoudt zich te | |
| | allen tijde het recht voor om af te zien van dit interview zonder opgave var | | |
| reden. | | | |
| | | Telefoonnr.: | <del></del> |
| - | Ik wil mee | | |
| Naa | m proefper | soon: | |
| Handtekening: | | | Datum :// |

| Proefpersoneninformatie | |
|---|---|
| Ik verklaar dat ik deze proefpersoon volledig heb geïnformeerd over het genoemde onderzoek. | |
| Als er tijdens het onderzoek informatie bekend wordt die de toestemming van de proefpersoon zou kunnen beïnvloeden, dan breng ik hem/haar daarvan tijdig op de hoogte. | |
| Naam onderzoeker (of diens vertegenwoordiger): | |
| Handtekening: | Datum: / / |
| <indien toepassing="" van=""></indien> | |
| Aanvullende informatie is gegeven door: | |
| Naam: | |
| Functie: | |
| Handtekening: | Datum: / / |

De proefpersoon krijgt een volledige informatiebrief mee, samen met een kopie van het getekende toestemmingsformulier.

<sup>\*</sup> Doorhalen wat niet van toepassing is.

## Bijlage D: toestemmingsformulier nabestaande

#### **MOSART-studie**

Een naaste van u neemt deel aan de MOSART-studie. Hij/zij heeft aangegeven toestemming te geven om na zijn/haar overlijden u te mogen benaderen voor een telefonisch interview door de onderzoeker over hoe u deze periode rond het overlijden ervaren hebt. Uiteraard benaderen wij u alleen hiervoor indien ook u hiervoor toestemming geeft.

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn voldoende beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen of te stoppen met het interview. Daarvoor hoef ik geen reden te geven.
- Ik weet dat sommige mensen mijn gegevens kunnen inzien. Die mensen staan vermeld in deze informatiebrief.
- Ik geef toestemming voor het verzamelen en gebruiken van mijn gegevens op de manier en voor de doelen die in de informatiebrief staan (zie ook sectie 4).
- Ik geef toestemming om mijn gegevens op de onderzoek-locatie nog 15 jaar na dit onderzoek te bewaren.
- Ik geef toestemming om de data die dit onderzoek oplevert eventueel in de toekomst te hergebruiken voor controle of verdere analyse in het kader van wetenschappelijk onderzoek.
- Ik wil meedoen aan dit interview.

| Naam nabestaande: | | | | |
|-------------------|-------|---|---|---|
| Handtekening: | Datum | : | / | / |

| Proefpersoneninformatie | |
|---|---|
| lk verklaar dat ik deze proefpersoon volledig heb geïnformeerd over het genoemde onderzoek. | |
| Als er tijdens het onderzoek informatie bekend wordt die de toestemming van de proefpersoon zou kunnen beïnvloeden, dan breng ik hem/haar daarvan tijdig op de hoogte. | |
| Naam onderzoeker (of diens vertegenwoordiger): | |
| • | Datum: / / |
| <pre><indien toepassing="" van=""></indien></pre> | |
| Aanvullende informatie is gegeven door: | |
| Naam: | |
| Functie: | |
| Handtekening: | Datum: / / |
| * Doorhalen wat niet van toenassing is | |

De nabestaande krijgt een volledige informatiebrief mee, samen met een kopie van het getekende toestemmingsformulier.

Doorhalen wat niet van toepassing is.